CLINICAL TRIAL: NCT01391663
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single and Multiple-Dose Study of the Pharmacokinetics and Pharmacodynamics of Alogliptin 12.5 mg, 25 mg and 50 mg in Healthy Korean Subjects
Brief Title: Pharmacokinetics and Pharmacodynamics Study of Alogliptin in Healthy Korean Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: SYR-322_106; U1111-1121-7268 (Registry Identifier: WHO)
Record Dates: First submitted 2011-07-08; First posted 2011-07-12 (Estimated); Results first posted 2013-03-22 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-02

CONDITIONS: Pharmacokinetics and Pharmacodynamics
Keywords: Drug Therapy
MeSH Terms: interventions — alogliptin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Alogliptin 12.5 mg QD (Experimental)
  Interventions: Drug: Alogliptin
- Alogliptin 25 mg QD (Experimental)
  Interventions: Drug: Alogliptin
- Alogliptin 50 mg QD (Experimental)
  Interventions: Drug: Alogliptin

INTERVENTIONS:
Drug: Alogliptin — Alogliptin 12.5 mg, tablets, orally, once daily for up to 7 days.
  Other Names: SYR-322
  Arms: Alogliptin 12.5 mg QD
Drug: Alogliptin — Alogliptin 25 mg, tablets, orally, once daily for up to 7 days.
  Other Names: SYR-322
  Arms: Alogliptin 25 mg QD
Drug: Alogliptin — Alogliptin 25 mg, tablets, orally, two tablets taken once daily for up to 7 days.
  Other Names: SYR-322
  Arms: Alogliptin 50 mg QD

SUMMARY:
The purpose of this study is to assess the Pharmacokinetics and Pharmacodynamics of alogliptin after a single or multiple administrations, once daily (QD), of oral alogliptin in healthy Korean subjects.

DETAILED DESCRIPTION:
Alogliptin is a selective, orally available inhibitor of dipeptidyl peptidase-4 being developed by Takeda Global Research & Development Center, Inc. as a treatment for type 2 diabetes mellitus. Inhibition of dipeptidyl peptidase-4 (DPP-4) prolongs the action of 2 important incretin hormones, glucagon-like peptide-1 (GLP-1) and glucose-dependent insulinotropic peptide (GIP). These hormones are responsible for increasing insulin synthesis, regulating β-cell proliferation, inhibiting gastric emptying and inhibiting glucagon secretion.

Evaluations of alogliptin and its clinical efficacy have been conducted in multiple countries including the United States and Japan. As development of alogliptin expands to other countries, additional studies are needed to bridge between the data previously acquired.

The main objective of this study is to assess the pharmacokinetics and pharmacodynamics of alogliptin in healthy Korean participants.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. The participant is a healthy adult male or female participant of Korean descent.
4. The participant is aged 18 to 55 years, inclusive, at the time of informed consent and first study medication dose.
5. The participant has a body mass index (BMI) between 18.0 and 26.0 kg/m2, inclusive at Screening.
6. A male participant who is non-sterilized and sexually active with a female partner of childbearing potential agrees to use adequate contraception from signing of informed consent throughout the duration of the study and for 12 weeks after last the dose.
7. A female participant of childbearing potential who is sexually active with a non-sterilized male partner agrees to use routinely adequate contraception from signing of informed consent throughout the duration of the study and for 30 days after the last dose of study drug.

Exclusion Criteria:

1. The participant has received any investigational compound within 30 days prior to Screening.
2. The participant has received alogliptin in a previous clinical study or as a therapeutic agent.
3. The participant is an immediate family member, study site employee, or in a dependant relationship with a study site employee who is involved in the conduct of this study (e.g., spouse, parent, child, sibling) or may consent under duress.
4. The participant has history of uncontrolled, clinically significant manifestations of metabolic (including diabetes mellitus, hypercholesterolemia, or dyslipidemia), endocrine, hematologic, pulmonary, cardiovascular, gastrointestinal, neurological, rheumatologic, skin and subcutaneous tissue disorders, infectious, hepatic, renal, urologic, immunologic, psychiatric or mood disorders (including any past history of suicide attempt), or a history of lactose intolerance, which may impact the ability of the participant to participate or potentially confound the study results.
5. Participant has a known hypersensitivity to any component of the formulation of alogliptin.
6. The participant has a positive urine drug result for drugs of abuse or alcohol at Screening or Check-in (Day -1).
7. The participant has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 1 year prior to the Screening visit or is unwilling to agree to abstain from alcohol and drugs throughout the study.
8. Participant has taken any excluded medication, supplements, or food products listed in the Excluded Medications and Dietary Products table.
9. If female, the participant is pregnant or lactating or intending to become pregnant before, during, or within 30 days after participating in this study; or intending to donate ova during such time period.
10. If male, the participant intends to donate sperm during the course of this study or for 12 weeks after the last dose.
11. Participant has evidence of current cardiovascular, central nervous system, hepatic, hematopoietic disease, renal dysfunction, metabolic or endocrine dysfunction, serious allergy, asthma hypoxemia, hypertension, seizures, or allergic skin rash. There is any finding in the participant's medical history, physical examination, or safety laboratory tests giving reasonable suspicion of a disease that would contraindicate taking alogliptin, or a similar drug in the same class, or that might interfere with the conduct of the study. This includes, but is not limited to, peptic ulcer disease, seizure disorders, and cardiac arrhythmias.
12. Participant has current or recent (within 6 months) gastrointestinal disease that would be expected to influence the absorption of drugs (i.e., a history of malabsorption, esophageal reflux, peptic ulcer disease, erosive esophagitis frequent [more than once per week] occurrence of heartburn, or any surgical intervention [e.g., cholecystectomy]).
13. Participant has a history of cancer, except basal cell carcinoma which has been in remission for at least 5 years prior to Day 1.
14. Participant has a positive test result for hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV), or a known history of human immunodeficiency virus infection at the Screening visit.
15. Participant has used nicotine-containing products (including but not limited to cigarettes, pipes, cigars, chewing tobacco, nicotine patch or nicotine gum) within 28 days prior to Check-in Day -1. Cotinine test is positive at Screening or Check-in (Day -1).
16. The participant has poor peripheral venous access.
17. Participant has donated or lost 450 mL or more of his or her blood volume (including plasmapheresis), or had a transfusion of any blood product within 30 days prior to Day 1.
18. Participant has a Screening or Check-in (Day -1) abnormal (clinically significant) electrocardiogram (ECG). Entry of any participant with an abnormal (not clinically significant) ECG must be approved, and documented by signature by the principal investigator.
19. Participant has abnormal Screening or Day -1 laboratory values that suggest a clinically significant underlying disease or participant with the following lab abnormalities: alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) >2x the upper limits of normal.
20. Participant has a hemoglobin value <12 g/dL at Screening only.
21. Participant has a systolic blood pressure ≥140 mm Hg or has a diastolic blood pressure ≥90 mm Hg at Screening or Check-in (Day -1).
22. Participant has a serum creatinine level >1.5 mg/dL at Screening only.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2011-07; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Director Clinical Science, Study Director — Takeda
Locations (1):
- Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at a single investigative site in South Korea from 25 July 2011 to 02 September 2011.
Pre-assignment Details: Healthy Korean participants were enrolled in either alogliptin 12.5 mg, 25 mg or 50 mg once-daily (QD) treatment groups.
Groups:
- Alogliptin 12.5 mg QD: Alogliptin 12.5 mg, tablets, orally, once daily for up to 7 days.
- Alogliptin 25 mg QD: Alogliptin 25 mg, tablets, orally, once daily for up to 7 days.
- Alogliptin 50 mg QD: Alogliptin 25 mg, tablets, orally, two tablets taken once daily for up to 7 days.
- Placebo: Placebo tablets, orally, two tablets taken once daily for up to 7 days.
Period: Overall Study
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Placebo
Started | 12 | 12 | 12 | 12
Completed | 12 | 12 | 11 | 12
Not Completed | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Placebo | Total
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 48
Age Continuous [Mean (Standard Deviation); unit: Years] | 26.6 (5.05) | 23.5 (2.75) | 25.3 (7.88) | 25.8 (2.17) | 25.3 (4.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 3 | 3 | 13
  Male | 8 | 9 | 9 | 9 | 35
Race/Ethnicity, Customized [Number; unit: participants]
  Korean | 12 | 12 | 12 | 12 | 48
  Other | 0 | 0 | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: cm] | 171.7 (9.05) | 170.3 (8.52) | 171.2 (8.62) | 168.9 (8.11) | 170.5 (8.37)
Weight [Mean (Standard Deviation); unit: kg] | 65.33 (8.76) | 63.37 (10.49) | 62.84 (9.78) | 60.85 (8.891) | 63.10 (9.34)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 22.17 (1.35) | 21.67 (2.31) | 21.53 (2.41) | 21.00 (1.525) | 21.59 (1.94)

OUTCOME MEASURES:

1. Primary Outcome: Cmax: Maximum Observed Plasma Concentration Pharmacokinetic Parameter
Description: Maximum observed plasma concentration (Cmax) is the peak plasma concentration after administrations of a single dose and multiple doses of the study drug
Time Frame: Day 1-4, Day 10
Population: Healthy Korean Participants
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 12
ng/mL
  Day 1 (n=12; n=12; n=12; n=12) | 55.28 (10.700) | 114.08 (36.611) | 246.00 (89.699) | NA (NA) — No values were collected for placebo Arm
  Day 10 (n=12; n=12; n=11; n=12) | 75.38 (14.708) | 154.83 (34.842) | 335.36 (61.983) | NA (NA) — No values were collected for placebo Arm

2. Primary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) Pharmacokinetic Parameter
Description: Time to reach the maximum plasma concentration (Tmax) after administrations of a single dose and multiple doses of the study drug
Time Frame: Day 1-4, Day 10.
Population: Healthy Korean Participants
Measure: Median (Full Range); unit: hr
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 12
hr
  Day 1 (n=12; n=12; n=12; n=12) | 1.49 [1.00 to 6.00] | 1.01 [0.52 to 3.033] | 3.00 [0.52 to 6.08] | NA [NA to NA] — No values were collected for placebo Arm
  Day 10 (n=12; n=12; n=11; n=12) | 1.02 [0.97 to 6.00] | 2.00 [0.98 to 6.00] | 1.02 [0.48 to 4.00] | NA [NA to NA] — No values were collected for placebo Arm

3. Primary Outcome: AUC(0-inf): Area Under the Plasma Concentration-time Curve From Time 0 to Infinity Pharmacokinetic Parameter
Description: Area under the plasma concentration-time curve from time 0 to infinity after administration of a single dose of the study drug.
Time Frame: Day 1-4
Population: Healthy Korean Participants
Measure: Mean (Standard Deviation); unit: ng·hr/mL
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 12
ng·hr/mL | 895.28 (78.639) | 1674.88 (308.115) | 3306.68 (530.295) | NA (NA) — No values were collected for placebo Arm

4. Primary Outcome: AUC(0-24): Area Under the Plasma Concentration-Time Curve From Time 0 to 24 Hours Pharmacokinetic Parameter.
Description: Area under the curve from 0 to 24 hours after administrations of a single dose and multiple doses of the study drug.
Time Frame: Day 1-4, Day 10.
Population: Healthy Korean Participants
Measure: Mean (Standard Deviation); unit: ng·hr/mL
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 12
ng·hr/mL
  Day 1 (n=12; n=12; n=12; n=12) | 601.65 (77.520) | 1174.76 (184.062) | 2488.48 (408.016) | NA (NA) — No values were collected for placebo Arm
  Day 10 (n=12; n=12; n=11; n=12) | 842.17 (84.110) | 1625.58 (397.301) | 3389.21 (406.082) | NA (NA) — No values were collected for placebo Arm

5. Primary Outcome: Terminal Phase Elimination Half-life (T1/2) Pharmacokinetic Parameter
Description: Time required for half of the drug to be eliminated from the plasma after administration of a single dose of the study drug.
Time Frame: Day 1-4
Population: Healthy Korean Participants
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 12
hr | 20.67 (2.067) | 19.45 (3.433) | 17.00 (3.104) | NA (NA) — No values were collected for placebo Arm

6. Primary Outcome: Oral Clearance (CL/F) Pharmacokinetic Parameter
Description: CL/F is apparent clearance of the drug from the plasma after administration of a single dose of the study drug.
Time Frame: Day 1-4
Population: Healthy Korean Participants
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 12
L/hr | 14.06 (1.241) | 15.30 (2.291) | 15.44 (2.214) | NA (NA) — No values were collected for placebo Arm

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) are adverse events (AEs) with an onset after the first dose of study drug (Day 1) and up to 30 ± 2 days after the last dose of study drug.
Description: An AE is defined as any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not it is considered related to the medicinal product.
Arm/Group | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Placebo
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 2/12 | 2/12 | 4/12 | 3/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alogliptin 12.5 mg QD (N=12) | Alogliptin 25 mg QD (N=12) | Alogliptin 50 mg QD (N=12) | Placebo (N=12)
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Headache (Nervous system disorders) | 1 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Epigastric Discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Feeling cold (General disorders) | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1
Thirst (General disorders) | 0 | 0 | 0 | 1
Tooth impacted (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Upper Respiratory Tract Infections (Infections and infestations) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be made without Sponsor's prior written approval. Any proposed publication or presentation will be submitted to Sponsor for review 60 days in advance of publication. Institution will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for an additional 60 days to preserve intellectual property.